CLINICAL TRIAL: NCT05814887
Title: Reduction of Mechanical IV Complication Using a New Medical Device
Acronym: ReLink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Peter Frykholm, Associate Professor, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ReLink
Record Dates: First submitted 2023-03-17; First posted 2023-04-18 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Catheter Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ReLink (Experimental): Medical device to be tested
  Interventions: Device: ReLink
- Control (No Intervention): Control, no medical device

INTERVENTIONS:
Device: ReLink — Medical device
  Arms: ReLink

SUMMARY:
Peripheral intravenous catheters are necessary for in-hospital medical treatment. Malfunction due to occlusion or dislodgement is common, and increases the burden on health care.

The aim of this study is to determine if the use of a new medical device has an impact on mechanical complications rate when peripheral intravenous (IV) catheter is used. The study will also investigate the safety, opinions of healthcare personnel and health economic effects of this new device,

DETAILED DESCRIPTION:
It is estimated that around 1.5 billion peripheral intravenous catheters (PIVC) are sold every year globally, and placing them is one of the most common invasive procedures in hospitalised patients, with up to 90% receiving one, yet there is a failure rate of up to 69%. Some of the most common causes of failure are considered to be phlebitis, subcutaneous infiltration, occlusion and dislodgement. These failure rates vary widely, where published data suggests rates of 8-44% for phlebitis, 5-21% for infiltration, 7.6-16% for occlusion and 5-10% for dislodgement. Phlebitis, commonly defined as an inflammatory process in the wall of a vein, resulting in a blood clot formation; while infiltration is defined as the inadvertent leakage of a solution into the surrounding tissue; occlusion is defined as PIVC failure due to blockage where flushing and/or aspiration is not possible, and dislodgement the complete accidental/inadvertent removal of the PIVC before intended. Previous studies have suggested that mechanical irritation could be an important factor resulting in PIVC failure. In the case of phlebitis, mechanical movements against the endothelial wall could initiate a cascade of prothrombotic events resulting in the formation of a blood clot, something that has been demonstrated in a simulated environment.

Therefore, there is a need to investigate potential new methods for prevention of these mechanical complications, and one way could be in the reduction of mechanical forces acting on the vessels. The aim of this study is to investigate the safety and effectiveness of a new medical device in reducing the number of mechanical complications during IV therapy.

The investigators have divided the research questions into a primary endpoint and secondary endpoints.

1. Primary endpoint:

   The rate of mechanical complications of an IV therapy session using a new medical device (ReLink) compared to using current 'state of the art'.
2. Secondary endpoint:

   * Frequency and severity of any adverse events
   * Healthcare workers opinion of the new medical device
   * The economic cost of these disruptions to the hospital or healthcare facility in terms of man-hours, and resources

The study is a randomized controlled trial to be run at Uppsala University Hospital. Patients will be randomly assigned to either the experimental group receiving IV infusion treatment using the new medical device ReLink, or the control group receiving IV infusion treatment without the device. Once the full intended IV infusion treatment has been completed, the same patient may be re-randomized and re-included in the trial. In case there is a mechanical complication resulting in the exchange of peripheral catheter, the patient will be re-randomized to either the control or intervention group. The risk of introducing a bias by re-randomizing the patients has been analysed and is considered to be minor. Firstly, in case of a re-randomization, this will take place after the follow-up of a peripheral catheter is completed. Secondly, re-randomization has been chosen instead of a cross-over design (where a patient's second peripheral catheter would automatically be selected to the other group) to avoid a spill-over effect from the patient themselves being biased against or in favour of using the device.

ELIGIBILITY:
Inclusion Criteria:

* The patient has or will get a PIVC expected to be used for continuous or intermittent IV infusion therapy. Continuous IV infusion is defined as an infusion ≥ 2h and intermittent as an infusion lasting 15min to < 2h.
* ≥18 years of age
* Speaks and understands Swedish

Exclusion Criteria:

* The PIVC is expected to be used for sampling only
* Pregnancy
* Unable to obtain informed consent or without an available Next-of-kin to provide surrogate informed consent
* Patients under palliative care
* Bolus IV infusion, defined as an infusion time of <15 min
* Phlebitis, infiltration or occlusion associated with PIVC that is already in place at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-05-04 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
The rate of mechanical complications of an IV therapy session using a new medical device (ReLink) compared to using current 'state of the art'. | Up to one week from randomization
  Mechanical complications is defined as phlebitis, subcutaneous infiltration, occlusion or dislodgement

SECONDARY OUTCOMES:
Frequency and severity of any adverse events | Up to one week from randomization
  Recording of any adverse events during the trial
Healthcare workers opinion of the new medical device | Within one week of removal of the device
  Questionnaire asking healthcare workers opinion, maximum score 5/ minimum score 0, high scores indicated better outcome
The economic cost of these disruptions to the hospital or healthcare facility in terms of man-hours, and resources | Through study completion, an average of 1 year
  Economical calculations based on additional materials and healthcare workers time

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, M.D., Ph.D., Principal Investigator — Dept of Anesthesia and Intensive Care, Uppsala University Hospital, 751 85 Uppsala, Sweden
Locations (1):
- Christopher Blacker, Uppsala, Uppsala County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blacker C, Modiri AR, Ljungman G, Frykholm P. The effects of a new device on mechanical complications of short peripheral intravenous catheters: A randomized controlled trial. J Vasc Access. 2025 Nov 11:11297298251389658. doi: 10.1177/11297298251389658. Online ahead of print. PMID 41216825